CLINICAL TRIAL: NCT00640575
Title: Subacromial Ultrasound-guided or Systemic Steroid Injection for Rotator Cuff Disease, a Randomized Double Blinded Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Ole Marius Ekeberg, University of Oslo
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sais-201204
Record Dates: First submitted 2008-03-09; First posted 2008-03-21 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2005-03

CONDITIONS: Rotator Cuff Disease
MeSH Terms: interventions — Triamcinolone; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Local
  Interventions: Drug: triamcinolone and lidocaine hydrochloride
- B (Active Comparator): Systemic
  Interventions: Drug: triamcinolone and lidocaine hydrochloride

INTERVENTIONS:
Drug: triamcinolone and lidocaine hydrochloride — Ultrasound-guided lidocaine hydrochloride 5 ml (10 mg/ml) injection in the subacromial bursa and a triamcinolone 2 ml (10 mg/ml) and 2 ml lidocaine hydrochloride (10 mg/ml) intramuscular injection in the gluteal region
  Other Names: Xyloacain (AstraZeneca); Kenakort-T (Bristol-Myers Squibb)
  Arms: B
Drug: triamcinolone and lidocaine hydrochloride — Ultrasound-guided injection of 2 ml triamcinolone (10 mg/ml) and 5 ml lidocaine hydrochloride (10 mg/ml) in the subacromial bursa and 4 ml intramuscular injection of lidocaine hydrochloride in the gluteal region
  Other Names: Kenacort-T (Bristol-Myers Squibb); Xylocain (AstraZeneca)
  Arms: A

SUMMARY:
Corticosteroid injections is a popular treatment option in shoulder disease. The evidence of effectiveness of corticosteroid injections is however contradicting. The importance of the accuracy of the steroid placement have been discussed and recently there are a few studies indicating better treatment effect if the injections are guided towards specific anatomical structures by real time ultrasound imaging. None of these studies have been double blinded. The aim of this study is to investigate the importance of placement of steroid injection in patients with rotator cuff disease by comparing systemic and ultrasound-guided injection in the subacromial bursa using a double blinded design.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years
* shoulder pain for more than 3 months
* pain at abduction of the affected shoulder
* less than 50 % reduced passive glenohumeral range of motion in no more than one direction of either abduction, external or internal rotation
* 2 of 3 positive isometric test of external rotation, internal rotation and abduction
* positive Hawkins-Kennedy impingement test

Exclusion Criteria:

* SPADI score below 30 points
* symptomatic acromioclavicular arthritis
* clinical and radiological findings indicating glenohumeral joint pathology
* referred pain from neck or internal organs
* clinical signs of a cervical syndrome
* generalized muscular pain syndrome with bilateral muscular pain in the neck and shoulders
* history of inflammatory arthritis
* diabetes mellitus type 1
* contraindications to local steroid or lidocaine hydrochloride injections
* corticosteroid injections last month before inclusion
* unable to respond to questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-03; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 2 and 6 weeks

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | 2 and 6 weeks
Pain in activity (7 point ordinal scale) | 2 and 6 weeks
Pain at rest (7 point ordinal scale) | 2 and 6 weeks
Change in main complaint (18 point ordinal scale) | 2 and 6 weeks
Active range of motion | 2 and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ole M Ekeberg, MD, Principal Investigator — University of Oslo

REFERENCES:
- [Derived] Ekeberg OM, Bautz-Holter E, Juel NG, Engebretsen K, Kvalheim S, Brox JI. Clinical, socio-demographic and radiological predictors of short-term outcome in rotator cuff disease. BMC Musculoskelet Disord. 2010 Oct 15;11:239. doi: 10.1186/1471-2474-11-239. PMID 20950433
- [Derived] Ekeberg OM, Bautz-Holter E, Tveita EK, Juel NG, Kvalheim S, Brox JI. Subacromial ultrasound guided or systemic steroid injection for rotator cuff disease: randomised double blind study. BMJ. 2009 Jan 23;338:a3112. doi: 10.1136/bmj.a3112. PMID 19168537